CLINICAL TRIAL: NCT05490771
Title: MATCH Treatment Subprotocol Z1F: Phase II Study of Copanlisib in Patients With Tumors With PIK3CA Mutations (PTEN Loss Allowed)
Brief Title: Testing Copanlisib as a Potential Targeted Treatment in Cancers With PIK3CA Mutations (MATCH-Subprotocol Z1F)
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2022-06209; NCI-2022-06209 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); EAY131-Z1F (Other: ECOG-ACRIN Cancer Research Group); EAY131-Z1F (Other: CTEP); U10CA180820 (NIH); U24CA196172 (NIH)
Record Dates: First submitted 2022-08-05; First posted 2022-08-08 (Actual); Results first posted 2023-02-28 (Actual); Last update posted 2025-11-14 (Actual); Status verified 2025-10

CONDITIONS: Advanced Lymphoma; Advanced Malignant Solid Neoplasm; Hematopoietic and Lymphatic System Neoplasm; Refractory Lymphoma; Refractory Malignant Solid Neoplasm; Refractory Multiple Myeloma
MeSH Terms: conditions — Lymphoma; Multiple Myeloma | interventions — Biopsy; copanlisib; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (copanlisib) (Experimental): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsies at screening and end of treatment and CT or MRI at baseline, every 2 cycles for the first 26 cycles, and then every 3 cycles thereafter until progressive disease or start of another MATCH treatment step.
  Interventions: Procedure: Biopsy Procedure; Procedure: Computed Tomography; Drug: Copanlisib Hydrochloride; Procedure: Magnetic Resonance Imaging

INTERVENTIONS:
Procedure: Biopsy Procedure — Undergo tumor biopsy
  Other Names: Biopsy; BIOPSY_TYPE; Bx
Procedure: Computed Tomography — Undergo CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Drug: Copanlisib Hydrochloride — Given IV
  Other Names: 5-Pyrimidinecarboxamide, 2-Amino-N-(2,3-dihydro-7-methoxy-8-(3-(4-morpholinyl)propoxy)imidazo(1,2-C)quinazolin-5-yl)-, Hydrochloride (1:2); Aliqopa; BAY 80-6946 Dihydrochloride; BAY-80-6946 Dihydrochloride; Copanlisib Dihydrochloride
Procedure: Magnetic Resonance Imaging — Undergo MRI
  Other Names: Magnetic Resonance; Magnetic Resonance Imaging (MRI); Magnetic resonance imaging (procedure); Magnetic Resonance Imaging Scan; Medical Imaging, Magnetic Resonance / Nuclear Magnetic Resonance; MR; MR Imaging; MRI; MRI Scan; MRIs; NMR Imaging; NMRI; Nuclear Magnetic Resonance Imaging; sMRI; Structural MRI

SUMMARY:
This phase II MATCH treatment trial identifies the effects of copanlisib hydrochloride (copanlisib) in patients whose cancer has a genetic change called PIK3CA mutation. Copanlisib may stop the growth of cancer cells by blocking PIK3, a protein needed for cell growth. Researchers hope to learn if copanlisib will shrink this type of cancer or stop its growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To evaluate the proportion of patients with objective response (OR) to targeted study agent(s) in patients with advanced refractory cancers/lymphomas/multiple myeloma.

SECONDARY OBJECTIVES:

I. To evaluate the proportion of patients alive and progression free at 6 months of treatment with targeted study agent in patients with advanced refractory cancers/lymphomas/multiple myeloma.

II. To evaluate time until death or disease progression. III. To identify potential predictive biomarkers beyond the genomic alteration by which treatment is assigned or resistance mechanisms using additional genomic, ribonucleic acid (RNA), protein and imaging-based assessment platforms.

IV. To assess whether radiomic phenotypes obtained from pre-treatment imaging and changes from pre- through post-therapy imaging can predict objective response and progression free survival and to evaluate the association between pre-treatment radiomic phenotypes and targeted gene mutation patterns of tumor biopsy specimens.

OUTLINE:

Patients receive copanlisib intravenously (IV) over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity. Patients also undergo tumor biopsies at screening and end of treatment and computed tomography (CT) or magnetic resonance imaging (MRI) at baseline, every 2 cycles for the first 26 cycles, and then every 3 cycles thereafter until progressive disease or start of another MATCH treatment step.

After completion of study treatment, patients are followed up every 3 months if less than 2 years from study entry, and then every 6 months for year 3 from study entry.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have met applicable eligibility criteria in the Master MATCH Protocol prior to registration to treatment subprotocol
* Patients must have PIK3CA mutation as determined via the MATCH Master Protocol
* Patients must have an electrocardiogram (ECG) within 8 weeks prior to treatment assignment and must have no clinically important abnormalities in rhythm, conduction or morphology of resting ECG (e.g. complete left bundle branch block, third degree heart block)
* Patients should stop using herbal medications at least 7 days prior to the first dose of copanlisib. Herbal medications include, but are not limited to: St. John's Wort, Kava, ephedra, gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, black cohosh and ginseng
* Patients with type I or II diabetes mellitus must have glycosylated hemoglobin A1c (HbA1c) =< 8.5% within 28 days from registration
* Absolute neutrophil count (ANC) >= 1.5 x 10^9 /L
* Platelets >= 100x10^9/L
* Hemoglobin (Hb) > 9 g/dl
* Total serum bilirubin < 2.0 mg/dL
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) < 2.5 x upper limit of normal (ULN) (< 5 x ULN in patients with liver metastases)
* Serum creatinine < 1.5 x ULN
* Men and women of child-bearing potential must agree to use contraception while receiving study treatment and for 1 month after the last dose of copanlisib

Exclusion Criteria:

* Patients must not have known hypersensitivity to copanlisib or compounds of similar chemical or biologic composition
* Patients must not have had prior therapy with copanlisib or other PI3K inhibitors, AKT inhibitors or mTOR inhibitors
* Patients must not have activating KRAS mutations
* Patients must not have HER2 positive (3+ by immunohistochemistry [IHC] or fluorescence in situ hybridization [FISH] ratio >= 2) breast cancer
* Patients must not have indolent non-Hodgkin lymphoma (NHL) (follicular lymphoma, small lymphocytic lymphoma [SLL]/chronic lymphocytic leukemia [CLL], lymphoplasmacytic lymphoma [LPL], marginal zone lymphoma) or DLBCL (diffuse large B cell lymphoma)
* Patients must not be on strong inhibitors or inducers of CYP3A4 within two weeks prior to start of study treatment and for the duration of study treatment
* Patients must not be on anti-arrhythmic therapy other than digoxin or beta-blockers
* Patients with non-healing wound, ulcer, or bone fracture are not eligible
* Patients with history of or current interstitial pneumonitis are not eligible

  * NOTE: For solid tumors, cytomegalovirus (CMV) polymerase chain reaction (PCR) can be obtained at the discretion of treating physician or local institutional guidelines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2018-06-20 (Actual); Primary Completion 2021-01-06 (Actual); Study Completion 2025-12-31 (Estimated)

CONTACTS AND LOCATIONS:
Overall Officials: Senthilkumar Damodaran, Principal Investigator — ECOG-ACRIN Cancer Research Group
Locations (1):
- ECOG-ACRIN Cancer Research Group, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subprotocol Z1F was activated on June 20, 2018. Thirty-five patients were enrolled between June 2018 and December 2018.
Pre-assignment Details: The PIK3CA mutations status was determined by a CLIA-approved assay performed in a NCI-MATCH approved laboratory for all patients in this arm. Mutation status was confirmed for 30 patients based on confirmation report as of August 1, 2019.
Groups:
- Treatment (Copanlisib): Patients receive copanlisib IV over 1 hour on days 1, 8, and 15 of each cycle. Cycles repeat every 28 days in the absence of disease progression or unacceptable toxicity
Period: Overall Study
Arm/Group | Treatment (Copanlisib)
Started | 35
Eligible | 31
Started Protocol Therapy | 30
Eligible and Treated | 28
Mutation Status Confirmed | 30
Eligible, Treated and Mutation Status Confirmed | 25
Completed | 0
Not Completed | 35
Not completed — Disease progression | 18
Not completed — Adverse Event | 3
Not completed — Other complicating disease | 1
Not completed — Withdrawal by Subject | 3
Not completed — Physician Decision | 1
Not completed — Still on treatment | 2
Not completed — Never start protocol therapy | 5
Not completed — Ineligible | 2

BASELINE CHARACTERISTICS:
Population: patients who were eligible, started protocol therapy, and had mutation status confirmed at the analysis time were the analyzable patients
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 25
Age, Continuous [Median (Full Range); unit: years] | 61 [42 to 78]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 9
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 22
  Unknown or Not Reported | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 1
  Black or African American | 2
  White | 21
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Response Rate (ORR)
Description: ORR is defined as the percentage of patients whose tumors have a complete or partial response to treatment among analyzable (ie, eligible, treated and PIK3CA mutation status confirmed) patients. Objective response is defined consistent with Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Details about how to define complete response and partial response can be found in the master protocol. 90% two-sided binomial exact confidence interval is calculated for ORR.
Time Frame: Tumor assessments occurred at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 30 months post registration
Population: Eligible, treated and PIK3CA mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 25
percentage of participants | 16 [6 to 33]
Statistical Analysis 1: Comparison: Treatment (Copanlisib); The ORR was compared against a null benchmark value of 5%. If the observed ORR were ≥5 of 31 (16%), it would then be concluded that the agent is promising and worthy of further investigation. When the number of analyzable cases (who were eligible and treated, and with outside assay results confirmed by the central MATCH assay) was <31, the one-sided exact binomial test would be used for significance test with one-side type I error rate of 5%; Test type: Superiority; p = 0.0341, one-sided exact binomial test

2. Secondary Outcome: 6-month Progression-Free Survival (PFS) Rate
Description: Progression-free survival is defined as time from treatment start date to date of progression or death from any cause, whichever occurs first.
  Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in NeuroOncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression. 6 month PFS rate was estimated using the Kaplan-Meier method, which can provide a point estimate for any specific time point.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles, and every 3 cycles thereafter until disease progression, up to 3 years post registration, from which 6-month PFS rate is determined
Population: Eligible, treated and PIK3CA mutation status confirmed
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 25
percentage of participants | 38 [22 to 53]

3. Secondary Outcome: Progression Free Survival (PFS)
Description: PFS was defined as time from treatment start date to date of disease progression or death from any causes, whichever occurred first.
  Median PFS was estimated using the Kaplan-Meier method. Disease progression was evaluated using the Response Evaluation Criteria in Solid Tumors version 1.1, the Cheson (2014) criteria for lymphoma patients, and the Response Assessment in Neuro-Oncology criteria for glioblastoma patients. Please refer to the protocol for detailed definitions of disease progression.
Time Frame: Assessed at baseline, then every 2 cycles for the first 26 cycles and every 3 cycles thereafter until disease progression, up to 3 years post registration
Population: Eligible, treated and PIK3CA mutation status confirmed
Measure: Median (90% Confidence Interval); unit: months
Arm/Group | Treatment (Copanlisib)
Number analyzed (Participants) | 25
months | 3.4 [1.8 to 6.6]

ADVERSE EVENTS:
Time Frame: Assessed every 28 days while on treatment and for 30 days after the end of treatment, up to 3 years post registration.
Description: All 35 patients enrolled in the trial were monitored for mortality, 30 of them started protocol therapy after registration and reported adverse events data. Serious adverse events are defined as grade 3 or higher adverse events.
Arm/Group | Treatment (Copanlisib)
All-Cause Mortality (participants affected / at risk) | 30/35
Serious Adverse Events (participants affected / at risk) | 17/30
Other Adverse Events (participants affected / at risk) | 27/30
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Copanlisib) (N=30)
Pruritus (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 1
Oral pain (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Meningitis (Infections and infestations) | 1
Alkaline phosphatase increased (Investigations) | 1
Weight loss (Investigations) | 1
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 8
Hypoglycemia (Metabolism and nutrition disorders) | 1
Hypophosphatemia (Metabolism and nutrition disorders) | 1
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Dizziness (Nervous system disorders) | 1
Syncope (Nervous system disorders) | 1
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Acute kidney injury (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 9
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Copanlisib) (N=30)
Anemia (Blood and lymphatic system disorders) | 7
Edema limbs (General disorders) | 2
Fatigue (General disorders) | 12
General disorders and administration site conditions - Other (General disorders) | 3
Pruritus (Skin and subcutaneous tissue disorders) | 3
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 8
Abdominal pain (Gastrointestinal disorders) | 3
Constipation (Gastrointestinal disorders) | 6
Diarrhea (Gastrointestinal disorders) | 11
Dry mouth (Gastrointestinal disorders) | 3
Gastroesophageal reflux disease (Gastrointestinal disorders) | 2
Mucositis oral (Gastrointestinal disorders) | 4
Nausea (Gastrointestinal disorders) | 10
Vomiting (Gastrointestinal disorders) | 4
Alkaline phosphatase increased (Investigations) | 2
Lymphocyte count decreased (Investigations) | 3
Neutrophil count decreased (Investigations) | 3
Platelet count decreased (Investigations) | 2
Weight loss (Investigations) | 4
White blood cell decreased (Investigations) | 3
Anorexia (Metabolism and nutrition disorders) | 5
Dehydration (Metabolism and nutrition disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 13
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypomagnesemia (Metabolism and nutrition disorders) | 3
Generalized muscle weakness (Musculoskeletal and connective tissue disorders) | 2
Musculoskeletal and connective tissue disorder - Other, spe (Musculoskeletal and connective tissue disorders) | 2
Dysgeusia (Nervous system disorders) | 4
Headache (Nervous system disorders) | 4
Blurred vision (Eye disorders) | 2
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2
Hypertension (Vascular disorders) | 6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (1):
  • Study Protocol (2019-08-12): https://cdn.clinicaltrials.gov/large-docs/71/NCT05490771/Prot_001.pdf